CLINICAL TRIAL: NCT02823769
Title: Clinical Evaluation of Restoration Made of SI-R21204 Resin Composite Based on S-PRG Filler Technology Versus Nano-hybrid Resin Composite: A Prospective Controlled Clinical Trial up to 3 Years
Brief Title: Clinical Evaluation of SI-R21204 Versus Nano-hybrid Resin Composite: A Prospective Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Shofu Inc. (Industry)
Responsible Party: Principal Investigator, Funda Ozturk Bozkurt, Prof.Dr., Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3215
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Caries
Keywords: clinical study; dental fillings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SI-R21204 resin composite (Experimental): Fillings made with a new dental filling material
  Interventions: Device: SI-R21204 resin composite
- Nanohybrid resin composite (Active Comparator): Fillings made with nanohybrid resin composite (Clearfil Majesty)
  Interventions: Device: Nanohybrid resin composite

INTERVENTIONS:
Device: SI-R21204 resin composite — Primary caries of posterior teeth will be restored using SI-R21204 resin composite. Procedures will be done under local anesthesia if necessary. The preperation and restoration of the tooth will be done according to to the guidelines for ordinary restorative techniques.
  Arms: SI-R21204 resin composite
Device: Nanohybrid resin composite — One of the cavities will be restored with a nanohybrid resin composite (Clearfil Majesty) as a control restoration wth ordinary restorative techniques.
  Arms: Nanohybrid resin composite

SUMMARY:
Despite the advances in adhesive restorative techniques and materials, dental caries still remains a critical concern even today. In addition, recurrent caries related to microleakage is a common mode of failure of directly placed resin composite restorations. Resin composites are particularly susceptible to recurrent caries due to polymerization contraction and also imperfect adhesion of restorative to tooth tissue. Thus, strong durable bond between adhesive restoratives and tooth tissue and increasing the resistance of teeth to acid by encouraging the development of remineralization are essential to withstand secondary caries. Fluoride has been documented as a major contributing factor for the decline in the incidence of dental caries and also it has been accepted as an agent in the prevention of caries. Giomers are a new group of anhydrous resin based direct adhesive restorative materials based on the filler technology (PRG) have both advantages of glass ionomers namely, fluoride release and recharge, and resin composites with excellent optical and mechanical properties. The chemistry of Giomer materials facilitates fluoride ion release with the potential for a lower incidence of recurrent caries that was accepted as a major factor to retreat a resin restoration. Limited number of studies is available on their fluoride release, and polishability, as well as clinical survival.

The objective of this controlled clinical trial is to evaluate the clinical performance of restorative material "SI-R21204 resin composite" versus a "nano-hybrid resin com-posite" materials for Class I and Class II cavities that needs to be restored in per-manent teeth.40 patients are recruited to the project which is carried out at the School of dentistry, Istanbul Medipol University, Turkey.

DETAILED DESCRIPTION:
The objective of this controlled clinical trial is to evaluate the clinical performance of restorative material "SI-R21204 resin composite" versus a "nano-hybrid resin com-posite" materials for Class I and Class II cavities that needs to be restored in per-manent teeth. Giomers are a new group of anhydrous resin based direct adhesive restorative materials based on the filler technology (PRG) to form a stable phase of glass ionomer in the restorative. These materials have both advantages of glass ionomers namely, fluoride release and recharge, and resin composites with excellent optical and mechanical properties. PRG fillers are fabricated by acid-base reaction of glass particles and polyacrylic acid in the presence of water and forms wet silicous hydrogel. S-PRG filler particles exhibit a three-layer structure where the glass core is enveloped by a stable glass-ionomer hydrogel. This hydrogel is surrounded by the "reforming phase," which provides structural protection for the hydrogel. These materials with S-PRG technology therefore, differ from polyacid modified composite resins because the glass ionomer hydrogel forms only after water uptake by the compomer resin matrix after polymerization. The chemistry of Giomer materials facilitates fluoride ion release with the potential for a lower incidence of recurrent caries that was accepted as a major factor to retreat a resin restoration. Limited number of studies is available on their fluoride release, and polishability, as well as clinical survival. The study will be carried out as a prospective study, with assessment of the restorationsafter three year.

The project includes 40 patients. Most of the patients have been recruited from the Istanbul Medipol University Dental Clinics in Istanbul. After giving their consent to take part in the study Class I & II restorations of both upper and lower molars and premolars are performed.The treatment procedure is: The patients are offered local anesthetic before treatment start. The cavity is excavated and filled according to the guidelines for composite restorations.

The control procedure is:

The restoration is evaluated according to marginal adaptation, cavo surface marginal discoloration, approximal contact, fractures, caries associated with restorations and postoperative hypersensitivity. The controls will take place after two weeks, one year, two years and three years.

ELIGIBILITY:
Inclusion Criteria:

* Primary caries removal
* Class I & II restorations
* No obvious untreated caries, dental health problems (regularly checked by a dentist)
* Good or moderate oral hygiene (plaque score of less than 30% in anterior region before treatment)
* No untreated periodontal disease (only DPSI 1, 2)
* Subjects had to present no active carious lesions
* Subjects had to be over the age of 18, be classified according to the American Society of Anesthesiologists (ASA) as ASA I or ASA II, present with good oral hy-giene, and be free of periodontal disease (probing depth and attachment levels within normal limits, no furcation involvement, and no mobility)
* Subjects had to agree to keep the scheduled recall appointments for data collec-tion and maintenance and plan to stay in the area for at least 3 years.

Exclusion Criteria:

* Composite or amalgam removal
* Caries extends cemento-enamel junction in Class II.
* Considerable horizontal and/or vertical mobility of teeth: tooth mobility index score 2 or 3
* Considerable periodontal disease without treatment (DPSI 3-, 3+ and 4)
* Endodontic treatment with extensive loss of tooth tissue
* Patients who still want to bleach their teeth or bleached teeth less than 3 weeks ago
* Excluding the teeth, with opposing natural dentition (either intact or restored with intracoronal or extracoronal fixed restorations), and with a minimum of 20 teeth
* Subjects who presented with severe wear facets and/or reported parafunctional activities such as clenching or nocturnal bruxism
* Subjects who were restored with a removable partial dental prosthesis (RPDP), unless the RPDP replaced the tooth that was planned to be restored in the study
* Subjects who were pregnant pregnant during the duration of the study
* Subjects who are known to be allergic to the ingredients of resin materials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04 (Actual); Study Completion 2020-08-16 (Actual)

PRIMARY OUTCOMES:
FDI (World Dental Federation) criteria for dental restorations assesment | 3 years
  2 independent evaluators The primary outcome will consist in the FDI (World Dental Federation) instrument for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010 . This instrument is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually.The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome. Hickel R, Peschke A, Tyas M, Mjör I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples.
  Clin Oral Investig. 2010 Aug;14(4):349-66.

SECONDARY OUTCOMES:
Plaque accumulation according to the Silness & Löe (1964) Plaque Index | 3 years
  [Time Frame: at 3 years] [Safety Issue: Yes] 0 = No plaque in the gingival area.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent
Gingival Inflammation according to the Silness & Löe (1964) Gingival Index. | 3 years
  0 = Normal gingival.
  1. = Mild inflammation-slight change in colour, slight oedema. No bleeding on probing
  2. = Moderate inflammation-redness, oedema and glazing. Bleeding on probing.
  3. = Severe inflammation-marked redness and oedema. Ulceration. Tendency to spontaneous bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Emir Yuzbasioglu, DDS,PhD, Principal Investigator — Medipol University; Mutlu Özcan, DDS,PhD, Principal Investigator — University of Zurich
Locations (1):
- Istanbul Medipol University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toz-Akalin T, Ozturk-Bozkurt F, Kusdemir M, Ozsoy A, Yuzbasioglu E, Ozcan M. Three-year clinical performance of direct restorations using low-shrinkage Giomer vs. nano-hybrid resin composite. Front Dent Med. 2024 Oct 9;5:1459473. doi: 10.3389/fdmed.2024.1459473. eCollection 2024. PMID 39917677